CLINICAL TRIAL: NCT01641952
Title: Non-interventional, Prospective, Multicenter Study to Assess Efficacy and Safety of MabtheRA (Rituximab) in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response or Intolerance to One Anti-TNF Agent - FAST 2 SWITCH Program
Brief Title: An Observational Study of MabThera/Rituxan (Rituximab) in Patients With Rheumatoid Arthritis and an Inadequate Response or Intolerance to One Anti-Tumor Necrosis Factor (Anti-TNF) Agent
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27953
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rituximab: Participants who had an inadequate response or intolerance to one anti- tumor necrosis factor (anti-TNF) agent received rituximab (Mabthera) at a dose determined by the investigator, guided by the recommendation in the Summary of Product Characteristics.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab at a dose determined by the investigator, guided by the recommendation in the Summary of Product Characteristics.
  Other Names: Mabthera

SUMMARY:
This observational, prospective, multicenter study will evaluate the efficacy and safety of MabThera/Rituxan in participants with active rheumatoid arthritis and an inadequate response or intolerance to one anti-TNF therapy. Participants who receive MabThera/Rituxan according to the current standard and in line with the summary of product characteristics at a dose of 1000 milligram (mg) intravenously on Days 1 and 15 will be followed for 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Participants with rheumatoid arthritis, eligible for treatment with MabThera/Rituxan in accordance with summary of product characteristics (SPC)
* Inadequate response to a single TNF inhibitor defined as change in disease activity score-28 erythrocyte sedimentation rate (DAS28-ESR) <1.2 or DAS28-ESR >3.5 at 5 months after first course of anti-TNF therapy
* Participants with a clinical and biological evaluation performed within 12 weeks prior to enrollment may be included

Exclusion Criteria:

* More than one previous anti-TNF therapies
* Any other biological therapy apart from the one anti-TNF therapy
* Hypersensitivity to rituximab or any of the excipients or to murine proteins
* Active severe infections
* Participants in a severely immunocompromised state
* Severe heart failure [New York Heart Association (NYHA) Class IV] or severe, uncontrolled cardiac disease
* Women of childbearing potential not willing to use contraception
* Pregnant or breastfeeding women
* Participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with active rheumatoid arthritis and an inadequate response or intolerant to one prior anti-TFN therapy initiated on treatment with MabThera/Rituxan
Sampling Method: Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2011-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Bucharest, Romania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 505 participants were recruited in 58 centers.
Period: Overall Study
Arm/Group | Rituximab
Started | 505
Treated | 504
Completed | 471
Not Completed | 34
Not completed — Lost to Follow-up | 28
Not completed — Adverse Event | 6

BASELINE CHARACTERISTICS:
Population: Full analysis population included all participants who has fulfilled the eligibility criteria, and signed the informed consent form, participated at the screening examination.
Arm/Group | Rituximab
Number analyzed (Participants) | 505
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.36 (10.681)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 434
  Male | 71

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participant With Good or Moderate Response According to European League Against Rheumatism (EULAR) Response Criteria
Description: The DAS28 score is a measure of the participant's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity], and ESR. DAS28 total scores range from 0 to 10. DAS28 <=3.2 indicates low disease activity, DAS28 >3.2 to 5.1 indicates moderate to high disease activity. A negative change from Baseline indicates improvement. The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline (CFB) and the level of disease activity reached. Good response: DAS28 <=3.2 and a CFB >1.2. Moderate response: DAS28 <=3.2 and CFB >0.6 to <=1.2, DAS28 >3.2 to <=5.1 and CFB >1.2 or >0.6 to <=1.2, DAS28 >5.1 and CFB >1.2. No response: DAS28 <=3.2 and CFB >=0.6, DAS28 >3.2 to <=5.1 and CFB <=0.6, DAS28 >5.1 and CFB >0.6 to <=1.2 or <=0.6.
Time Frame: Week 20
Population: Full analysis population included all participants who has fulfilled the eligibility criteria, and signed the informed consent form, participated at the screening examination. Here, number of participants analyzed is the participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 488
percentage of participants
  Present <=3.2; CFB >1.2 | 0
  Present <=3.2; CFB >0.6 to <=1.2 | 8.20
  Present >3.2 to <=5.1; CFB >1.2 | 43.03
  Present >3.2 to <=5.1; CFB >0.6 to <=1.2 | 9.00
  Present >5.1; CFB >1.2 | 14.54

2. Primary Outcome: Change From Baseline in DAS28-ESR at Week 20
Description: DAS28 was calculated from SJC and TJC using an assessment of 28 joints, the erythrocyte sedimentation rate (ESR) (milliliter per hour [ml/hr]), and Patient's Global Assessment (PGH) of disease activity [measured on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS) where 0=no disease activity and 100=worst disease activity]. DAS28 was calculated using the following formula: DAS28 = 0.56*square root (sqrt) (TJC28) + 0.28*sqrt(SJC28) + 0.70*natural logarithm (ln) (ESR) + 0.014*PGH of disease activity. Total score range: 0-10, with a higher score indicated more disease activity. DAS28 <=3.2 implied low disease activity, DAS >3.2 to 5.1 implied moderate disease activity and DAS >5.1 implied high disease activity, and DAS28 <2.6 = clinical remission.
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 489
units on a scale | -1.53458 [-1.66 to -1.40]

3. Primary Outcome: Mean DAS28-ESR Score at Visit 4 (Week 20)
Description: DAS28 was calculated from SJC and TJC using an assessment of 28 joints, the erythrocyte sedimentation rate (ESR) (milliliter per hour [ml/hr]), and Patient's Global Assessment (PGH) of disease activity (measured on a 0 to 100 mm Visual Analogue Scale [VAS] where 0=no disease activity and 100=worst disease activity). DAS28 was calculated using the following formula: DAS28 = 0.56*square root (sqrt) (TJC28) + 0.28*sqrt(SJC28) + 0.70*natural logarithm (ln) (ESR) + 0.014*PGH of disease activity. Total score range: 0-10, with a higher score indicated more disease activity. DAS28 <=3.2 implied low disease activity, DAS >3.2 to 5.1 implied moderate disease activity and DAS >5.1 implied high disease activity, and DAS28 <2.6 = clinical remission.
Time Frame: Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 488
units on a scale | 3.8218 (1.26061)

4. Primary Outcome: Percentage of Participants With Change in DAS28-ESR of Greater Than or Equal (>=) 1.2 After First Course of Treatment
Description: as for outcome 3
Time Frame: Week 20
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 488
percentage of participants | 57.99

5. Primary Outcome: Percentage of Participants With EULAR Response
Description: The DAS28 score is a measure of the participant's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity], and ESR. DAS28 total scores range from 0 to 10. DAS28 <=3.2 indicates low disease activity, DAS28 >3.2 to 5.1 indicates moderate to high disease activity. A negative CFB indicates improvement. The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of CFB and the level of disease activity reached. Good response: DAS28 <=3.2 and a CFB >1.2. Moderate response: DAS28 <=3.2 and CFB >0.6 to <=1.2, DAS28 >3.2 to <=5.1 and CFB >1.2 or >0.6 to <=1.2, DAS28 >5.1 and CFB >1.2. No response: DAS28 <=3.2 and CFB >=0.6, DAS28 >3.2 to <=5.1 and CFB <=0.6, DAS28 >5.1 and CFB >0.6 to <=1.2 or <=0.6.
Time Frame: Week 20
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 488
percentage of participants
  Present <=3.2; CFB>1.2 | 0
  Present <=3.2; CFB>0.6 to <=1.2 | 8.20
  Present <=3.2; CFB <=0.6 | 17.62
  Present >3.2 to <=5.1; CFB >1.2 | 43.03
  Present >3.2 to <=5.1; CFB >0.6 and <=1.2 | 9.00
  Present >3.2 to <=5.1; CFB <=0.6 | 0
  Present >5.1; CFB >1.2 | 14.54
  Present >5.1; CFB >0.6 to <=1.2 | 0
  Present >5.1; CFB <=0.6 | 0
  No improvement | 8

6. Primary Outcome: Percentage of Participants With EULAR Response in Subgroup of Participants Who Had Been Treated With Anti-TNF Previously
Description: as for outcome 5
Time Frame: Week 20
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 488
percentage of participants
  No treatment; DAS 28 >3.2 to <=5.1 | 0
  No treatment; DAS 28 >5.1 | 0.83
  Actemra; DAS 28 >3.2 to <=5.1 | 0
  Actemra; DAS 28 >5.1 | 4.16
  Certolizumab; DAS 28 >3.2 to <=5.1 | 0
  Certolizumab; DAS 28 >5.1 | 0.83
  Golimumab; DAS 28 >3.2 to <=5.1 | 0
  Golimumab; DAS 28 >5.1 | 10
  Rituximab; DAS 28 >3.2 to <=5.1 | 0
  Rituximab; DAS 28 >5.1 | 3.33
  Tocilizumab; DAS 28 >3.2 to <=5.1 | 40.83
  Tocilizumab; DAS 28 >5.1 | 40

7. Primary Outcome: Percentage of Participants With Remission (DAS28 <2.6) and Low Disease Activity Following Each Treatment Course
Description: as for outcome 3
Time Frame: Week 20
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 488
percentage of participants
  Remission (DAS28 <2.6) | 16.19
  Low Disease Activity | 15

8. Primary Outcome: Number of Participants With Remission (DAS28 <2.6) and Low Disease Activity Following Each Treatment Course for Subgroup of Participants Who Had Been Treated With Etanercept or Adalimumab or Infliximab Before Rituximab
Description: The DAS28 score is a measure of the participant's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity], and ESR. DAS28 total scores range from 0 to 10. DAS28 <=3.2 indicates low disease activity, DAS28 >3.2 to 5.1 indicates moderate to high disease activity. A negative change from Baseline (CFB) indicates improvement. The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of CFB and the level of disease activity reached. Good response: DAS28 <=3.2 and a CFB >1.2. Moderate response: DAS28 <=3.2 and CFB >0.6 to <=1.2, DAS28 >3.2 to <=5.1 and CFB >1.2 or >0.6 to <=1.2, DAS28 >5.1 and CFB >1.2. No response: DAS28 <=3.2 and CFB >=0.6, DAS28 >3.2 to <=5.1 and CFB <=0.6, DAS28 >5.1 and CFB >0.6 to <=1.2 or <=0.6.
Time Frame: Week 20
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 488
participants
  Adalimumab | 18
  Etanercept | 18
  Infliximab | 24

9. Primary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to 39 months
Population: Safety population included all participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 504
participants | 16

10. Secondary Outcome: Health Assessment Questionnaire (HAQ) Score at Week 20
Description: HAQ is a self-completed patient questionnaire specific for rheumatoid arthritis (RA). It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities. Each domain has at least 2 component questions. There are 4 possible responses for each component 0=without any difficulty 1=with some difficulty 2=with much difficulty 3=unable to do. Calculate HAQ the patient must have a domain score for at least 6 of 8 domains. The HAQ is the sum of the scores, divided by the number of domains that have a score (in range 6-8) for a total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from baseline indicated improvement.
Time Frame: Baseline and Week 20
Population: Intent to treat population included all participants who has fulfilled the eligibility criteria, and signed the informed consent form, participated to the screening exam, and have completed the baseline visit and at least one further assessment. Here, number of participant analysed is the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 488
units on a scale
  Baseline | 2.62 (0.737)
  Week 20 | 1.85 (0.715)

ADVERSE EVENTS:
Time Frame: up to 39 months
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 14/504
Other Adverse Events (participants affected / at risk) | 3/504
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=504)
Hypothermia (Injury, poisoning and procedural complications) | 1
Accelerated hypertension (Vascular disorders) | 1
Blood triglycerides increased (Metabolism and nutrition disorders) | 1
Peripheral venous disease (Vascular disorders) | 2
Parkinson Diseases (Nervous system disorders) | 1
Leg amputation (Surgical and medical procedures) | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1
Brain abscess (Infections and infestations) | 1
Oral cavity cancer metastatic (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Systemic inflammatory response syndrome (Immune system disorders) | 1
Influenza (Infections and infestations) | 1
Instillation site urticaria (Injury, poisoning and procedural complications) | 2
Anaphylactic shock (Immune system disorders) | 1
Seizure (Nervous system disorders) | 1
Pulmonary tuberculosis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=504)
Blood iron decreased (Investigations) | 1
Chronic gastritis (Immune system disorders) | 1
Tooth abscess (Infections and infestations) | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.